CLINICAL TRIAL: NCT04365933
Title: A Phase 2a Open-label Study of the Oral Farnesoid X Receptor (FXR) Modulator EYP001a to Assess Its Safety and Anti-viral Effect in Chronic Hepatitis B (CHB) Patients in Combination With Pegylated Interferon alpha2a (Peg-IFN) Alone and With Entecavir (ETV)
Brief Title: A Study of the Oral Farnesoid X Receptor Modulator EYP001a to Assess Its Safety and Anti-viral Effect in Chronic Hepatitis B Patients in Combination With Pegylated Interferon alpha2a Alone and With Entecavir
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Enyo Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EYP001-203
Record Dates: First submitted 2020-04-23; First posted 2020-04-28 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): EYP001a Dose A QD + ETV 0.5 mg QD + peg-IFN dosed per body surface area (180 µg, 135 µg or 90 µg) QW
  Interventions: Drug: EYP001a; Drug: Entecavir; Drug: Pegylated interferon alpha2a
- Arm 2 (Experimental): EYP001a Dose A QD + peg-IFN dosed per body surface area (180 µg, 135 µg or 90 µg) QW
  Interventions: Drug: EYP001a; Drug: Pegylated interferon alpha2a

INTERVENTIONS:
Drug: EYP001a — Oral tablets
Drug: Entecavir — Oral tablets
  Arms: Arm 1
Drug: Pegylated interferon alpha2a — Subcutaneous

SUMMARY:
This is a multi centre, two parallel arm, randomized, open-label, Phase 2a experimental study of oral Farnesoid X Receptor (FXR) modulator EYP001a to assess its safety and anti-viral effect when administered to non-treated (treatment naive or off treatment) chronic Hepatitis B (CHB) patients in combination with entecavir (ETV) and pegylated interferon alpha2a (peg-IFN). An experimental treatment period of 16 weeks will be followed by a 24 week maintenance period with ETV standard of care (SoC).

DETAILED DESCRIPTION:
In total 30 eligible patients will be enrolled and randomized at approximately 7 study sites.

Patients will be randomized prior to study drug (EYP001a, ETV and peg-IFN) administration on Day 1 in the ratio of 1:1 into 2 treatment arms:

* Arm 1: EYP001a QD + ETV 0.5 mg QD + peg-IFN dosed per body surface area (180 µg, 135 µg or 90 µg) QW (± 3 days) (15 patients)
* Arm 2: EYP001a QD + peg-IFN dosed per body surface area (180 µg, 135 µg or 90 µg) QW (± 3 days) (15 patients)

Patients enrolled in the study will be assessed as outpatients. Patient screening will occur no more than 37 days prior to the Day 1 visit. Eligible patients will undergo further assessments on Day 1 to qualify for study drug administration on Day 1.

The visits during the study are planned as below:

* Screening visit: 5 weeks (37 days)
* 16 weeks treatment period
* 24 weeks maintenance period. During maintenance period patients are kept on ETV until the end of the trial at Week 40.

ELIGIBILITY:
Inclusion Criteria:

* Has given voluntary written informed consent before performance of any study related procedure.
* Are treatment naive or without HBV treatment for at least 60 days or 5 times the elimination half-life, whichever is longer.
* Patient has CHB:

  1. HBV DNA ≥ 20,000 IU/mL for HBeAg positive and ≥2'000 for HBeAg negative and
  2. HBsAg ≥ 2.5 log10 IU/mL.
* Has liver imaging to screen for hepatocellular carcinoma or concomitant pancreaticobiliary disease either in the prior 6 months or at screening.
* Patient is not of childbearing potential or, if of childbearing potential, is not pregnant as confirmed by a negative serum human chorionic gonadotropin test at screening and is not planning a pregnancy during the course of the study.

Exclusion Criteria:

* Is an employee of a clinical research organization, vendor, or Sponsor involved with this study.
* Has known hepatocellular carcinoma or pancreaticobiliary disease.
* Neutropenia (defined by two confirmed values during Screening period of < 1500/μL).
* Has Gilbert syndrome.
* Shows evidence of worsening liver tests, defined as either a confirmed (2 assessments at least 3 days apart) increase > 2 ULN ALT or AST or an increase of > 1.5 × baseline value of TBL or associated with clinical signs or symptoms of liver impairment.
* Has known or suspected non-CHB liver disease
* History of cirrhosis or liver decompensation, including ascites, hepatic encephalopathy, or presence of oesophageal varices.
* Probable or possible F4 stage with a vibration controlled transient elastography (VCTE) > 11.7 kPa leads to exclusion
* Has known history of alcohol abuse or daily heavy alcohol consumption
* Has any of the following exclusionary laboratory results at screening:

  1. ALT > 2 × ULN, AST > 2 × ULN
  2. INR > 1.2 × ULN, (normal range is 0.8 to 1.2)
  3. Platelet count < 100 G/L
  4. Estimated glomerular filtration rate < 50 mL/min/1.73m2 (the Modification of Diet in Renal Disease formula)
  5. Thyroid-stimulating hormone > 1.5 × ULN or abnormal free triiodothyronine or free thyroxine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
Number of Treatment-emergent adverse events | 16 weeks
  Number of Treatment-emergent adverse events including serious adverse events
Measurement of HBsAg decline | 16 weeks
  Measurement of HBsAg decline (Δ log10) from Day 1 to Week 16 of treatment period

SECONDARY OUTCOMES:
Measurement of HBsAg decline | 40 weeks
  Measurement of HBsAg decline (Δ log10)
Measurement of HBV-DNA decline | 40 weeks
  Measurement of HBV-DNA decline (Δ log10)
Measurement of HBV-pgRNA decline | 40 weeks
  Measurement of HBV-pgRNA decline (Δ log10)
Measurement of HBcrAg decline | 40 weeks
  Measurement of HBcrAg decline (Δ log10)
Concentration of EYP001a - Pharmacokinetic | 20 weeks
  Assessment of fasted plasma concentrations of EYP001a or any active metabolites using a validated liquid chromatography-mass spectrometry
Concentration of C4 - Pharmacodynamic biomarker | 40 weeks
  Assessment of concentrations of plasma C4 (7α hydroxy 4 cholesten 3 one)
Concentration of FGF19 - Pharmacodynamic biomarker | 40 weeks
  Assessment of concentrations of plasma FGF19 over time (Fibroblast Growth Factor 19)
Concentration of Bile Acids - Pharmacodynamic biomarker | 40 weeks
  Assessment of concentrations over time of plasma Bile Acids (chenodeoxycholic acid, deoxycholic acid, lithocholic acid)

CONTACTS AND LOCATIONS:
Locations (6):
- ENYO PHARMA Investigative site HK01, Hong Kong, Hong Kong
- ENYO PHARMA Investigative site KR01, Busan, South Korea
- Taiwan (4):
  - ENYO PHARMA Investigative site TW03, Kaohsiung City
  - ENYO PHARMA Investigative site TW04, Kaohsiung City
  - ENYO PHARMA Investigative site TW01, Taipei
  - ENYO PHARMA Investigative site TW02, Taoyuan District

IPD SHARING:
Plan to Share IPD: No